CLINICAL TRIAL: NCT02940106
Title: Investigation of the Clinical Pregnancies Obtained After Cryopreservation of Donor Oocytes With an Open or Closed Device
Brief Title: Clinical Pregnancies After Cryopreservation of Donor Oocytes With an Open or Closed Device
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: enrollment too slow, too many variables included in the study
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Neelke De Munck, Master in Science, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2016/245
Record Dates: First submitted 2016-10-11; First posted 2016-10-20 (Estimated); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Infertility
Keywords: oocyte cryopreservation; closed vitrification; open vitrification
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- closed device (Placebo Comparator): Standard cryopreservation system.
  Interventions: Device: CBSvit device
- open device (Active Comparator): New cryopreservation system.
  Interventions: Device: Cryotop device

INTERVENTIONS:
Device: Cryotop device — a different device for oocyte vitrification (with a very high cooling rate)
  Other Names: Cryotop open vitrification device (Kitazato)
  Arms: open device
Device: CBSvit device — a different device for oocyte vitrification (with a lower cooling rate)
  Other Names: CBSvit closed vitrification device (CryoBioSystems vitrification device)
  Arms: closed device

SUMMARY:
This randomized pilot study will assess if there is a difference in clinical pregnancies using donor oocytes cryopreserved in either a closed or a semi-closed vitrification device.

DETAILED DESCRIPTION:
Oocyte cryopreservation was optimized by the use of a new technique: vitrification. Vitrification can be performed using either open devices (where the oocytes are in direct contact with the liquid nitrogen) or closed systems (where the oocytes are never in contact with liquid nitrogen). Previous studies have associated the use of open devices to higher oocyte survival rates and better embryo development. However, any beneficial effect on clinical pregnancy rates is yet to be proven. Hence, the objective of this study is to compare the clinical pregnancy rates of open and closed oocyte vitrification devices.

ELIGIBILITY:
Inclusion Criteria:

* this is a pragmatic randomized clinical trial. Hence, all consenting oocyte recipients will be eligible for the study

Exclusion Criteria:

* women who do not consent or that cannot comprehend the investigational nature of the study

Ages: 18 Years to 47 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy | 7 weeks
  Pregnancy determined by ultrasound

SECONDARY OUTCOMES:
survival | 1 week
  oocyte survival post-warming based on the morphological appearance of the oocytes immediately after warming: degenerated oocytes are non-surviving oocytes; oocytes with a normal morphological appearance are surviving oocytes
fertilization | 1 week
  oocyte fertilization post-insemination: the day after oocyte insemination fertilization is checked: if one male and one female pronucleus appear, the oocyte is fertilized. if both nuclei are not present or more nuclei are present, the oocyte is considered not fertilized.
embryo development | 2 weeks
  embryo development post-fertilization: on day 3 of pre-implantation development, the embryo is scored for the number of cells, fragmentation, appearance of nuclei and other embryological parameters: based on these parameters, an embryological score is given to the embryo. On day 5 of development (blastocyst stage) another score is given to the embryo based on the appearance of the trophectoderm and inner cell mass cells.

CONTACTS AND LOCATIONS:
Overall Officials: Neelke De Munck, MSc., Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] De Munck N, Santos-Ribeiro S, Stoop D, Van de Velde H, Verheyen G. Open versus closed oocyte vitrification in an oocyte donation programme: a prospective randomized sibling oocyte study. Hum Reprod. 2016 Feb;31(2):377-84. doi: 10.1093/humrep/dev321. Epub 2016 Jan 2. PMID 26724798